CLINICAL TRIAL: NCT02747953
Title: An Open Label Compassionate Use Programme of Gilotrif (Afatinib) in Advanced Non-Small Cell Lung Cancer Patients Pre-treated With Erlotinib or Gefitinib
Brief Title: Gilotrif (Afatinib) in Advanced Non-Small Cell Lung Cancer Patients Pre-treated With Erlotinib or Gefitinib
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Keunchil Park, Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-09-011
Record Dates: First submitted 2013-10-22; First posted 2016-04-22 (Estimated); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Afatinib

ARMS (1):
- afatinib (Experimental)
  Interventions: Drug: Gilotrif

INTERVENTIONS:
Drug: Gilotrif — 50 mg with an option to reduce the dose to 40mg or 30 mg once a day Continuous daily dosing, one course consists of 28 days. Patients are eligible for repeated treatment courses in the absence of disease progression and undue toxicity.
  Other Names: Afatinib

SUMMARY:
The program will provide early access to the investigational drug gilotrif in patients with advanced non-small cell lung cancer who have failed at least 6 months on erlotinib or gefitinib.

The Compassionate Use Programme will also provide additional safety information on gilotrif use.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with pathologically confirmed diagnosis of adenocarcinoma of the lung Stage IV with progressive disease following at least one line of platinum-based cytotoxic chemotherapy
2. Patients progressing after clinical benefit on erlotinib or gefitinib: clinical benefit is defined as stable disease for at least 6 months, or a complete or partial response, or the presence of an activating mutation of the epidermal growth factor (EGF) receptor family.
3. No further treatment option is available.
4. Male and female patients age ≥18 years.
5. Written informed consent that is consistent with International Conference on Harmonisation-Good Clinical Practice (ICH-GCP) guidelines and local law.

Exclusion Criteria:

1. Significant or recent acute gastrointestinal disorders with diarrhoea as a major symptom.
2. Patients who have any other life-threatening illness or organ system dysfunction, which in the opinion of the investigator, would compromise patient safety.
3. History of cardiac disease that is clinically significant, as judged by the investigator or uncontrolled cardiac disease (including congestive heart failure, angina, myocardial infarction, arrhythmia, including New York Heart Association (NYHA) functional classification of 3).
4. Aspartate amino transferase (AST) or alanine amino transferase (ALT) ≥ three times the upper limit of normal (if related to liver metastases ≥ five times the upper limit of normal).
5. Bilirubin ≥1.5 mg/dl
6. Serum creatinine ≥ 1.5 times of the upper normal limit or calculated/measured creatine clearance ≤ 45ml/min
7. Women of child-bearing potential or men who are able to father a child unwilling to use a medically acceptable method of contraception during the treatment.
8. Pregnancy or breast feeding.
9. Pre-existing Interstitial Lung Disease (ILD).
10. Patients suitable to be included into afatinib clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-07; Primary Completion 2014-12 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
response rate | 6 months